CLINICAL TRIAL: NCT02713386
Title: A Phase I/II Study of Ruxolitinib With Front-Line Neoadjuvant and Post-Surgical Therapy in Patients With Advanced Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Ruxolitinib Phosphate, Paclitaxel, and Carboplatin in Treating Patients With Stage III-IV Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GY007; NCI-2016-00203 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY007; NRG-GY007 (Other: NRG Oncology); NRG-GY007 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2024-10-24 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube High Grade Serous Adenocarcinoma; FIGO Stage III Ovarian Cancer 2014; FIGO Stage IIIA Ovarian Cancer 2014; FIGO Stage IIIA1 Ovarian Cancer; FIGO Stage IIIA2 Ovarian Cancer; FIGO Stage IIIB Ovarian Cancer 2014; FIGO Stage IIIC Ovarian Cancer 2014; FIGO Stage IVA Ovarian Cancer 2014; FIGO Stage IVB Ovarian Cancer 2014; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian High Grade Serous Adenocarcinoma; Primary Peritoneal Endometrioid Adenocarcinoma; Primary Peritoneal High Grade Serous Adenocarcinoma; Stage III Fallopian Tube Cancer AJCC v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Carboplatin; Paclitaxel; Taxes; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (paclitaxel and carboplatin) (Active Comparator): See Detailed Description.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Procedure: Therapeutic Conventional Surgery
- Arm II (ruxolitinib, paclitaxel, and carboplatin) (Experimental): See Detailed Description.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Ruxolitinib Phosphate; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi; Jakavi
  Arms: Arm II (ruxolitinib, paclitaxel, and carboplatin)
Procedure: Therapeutic Conventional Surgery — Undergo TRS

SUMMARY:
This phase I/II trial studies the side effects and the best dose of ruxolitinib phosphate when given together with paclitaxel and carboplatin and to see how well they work in treating patients with stage III-IV epithelial ovarian, fallopian tube, or primary peritoneal cancer. Ruxolitinib phosphate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ruxolitinib phosphate together with paclitaxel and carboplatin may be a better treatment for epithelial ovarian, fallopian tube, or primary peritoneal cancer compared to paclitaxel and carboplatin alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether treatment with ruxolitinib phosphate (ruxolitinib) in combination with conventional neoadjuvant and post-surgical chemotherapy is safe and tolerable in the primary therapy for epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. (Phase I) II. Demonstrate whether treatment with ruxolitinib in combination with conventional neoadjuvant and post-surgical chemotherapy results in a prolonged progression-free survival when compared to chemotherapy alone, in primary therapy for epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. (Phase II)

SECONDARY OBJECTIVES:

I. Determine frequency of patients who do not receive surgery within 6 weeks of completing cycle 3 therapy for reasons other than non-response, disease progression, or medical contraindications. (Phase I) II. Determine if continuation of ruxolitinib as maintenance therapy in participants who complete 6 cycles of standard chemotherapy in combination with ruxolitinib and have not experienced unacceptable toxicity or disease progression is safe and tolerable. (Phase I) III. Determine the impact of ruxolitinib in combination with chemotherapy on progression-free survival as a function of proposed exploratory biomarkers - ALDH+ CD133+ (possibly also CD24+ CK19+) co-staining by AQUA immunofluorescence (IF); ratio of tumor expression of CD8:FOXP3 by immunohistochemistry (IHC); and tumor CD3, CD4, TAI-1, HLA class I and II, CD68 expression by IHC in archived tumor tissue, BRCA status, and serum C-reactive protein (CRP) and IL-6 levels in pre-treatment serum. (Phase II) IV. Investigate the prognostic significance of exploratory laboratory parameters in terms of both progression-free survival and overall survival in women receiving conventional chemotherapy alone. (Phase II) V. Determine whether treatment with ruxolitinib in combination with conventional chemotherapy is associated with total gross resection rate at time of interval cytoreductive surgery. (Phase II) VI. Determine whether treatment with ruxolitinib in combination with conventional chemotherapy is associated with complete pathologic response defined at interval cytoreductive surgery. (Phase II) VII. Demonstrate whether treatment with ruxolitinib in combination with conventional chemotherapy results in an improvement in overall survival in primary management of epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of ruxolitinib phosphate, followed by a phase II study.

PHASE I PORTION OF STUDY IS COMPLETE (04/06/2018)

PHASE I (CYCLES 1-3): Patients receive ruxolitinib phosphate orally (PO) twice daily (BID) on days 1-21, paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Within 6 weeks after completion of cycle 3, patients undergo tumor reductive surgery (TRS).

PHASE I (CYCLES 4-6): Within 6 weeks of TRS, patients receive ruxolitinib phosphate PO BID on days 1-21, paclitaxel IV over 1 hour on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. If TRS is not performed due to non-response or medical contraindications and criteria for discontinuation of protocol therapy have not been met, patients should resume ruxolitinib phosphate, paclitaxel, and carboplatin within 6 weeks of completing cycle 3 of therapy.

MAINTENANCE THERAPY: Within 3 weeks after completion of cycle 6, patients receive ruxolitinib phosphate PO BID. Treatment continues in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I (CYCLES 1-3): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Within 6 weeks after completion of cycle 3, patients undergo TRS.

ARM I (CYCLES 4-6): Within 4 weeks of surgery (or within 6 weeks of completion of cycle 3 in patients who do not undergo TRS), patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity.

ARM II (CYCLES 1-3): Patients receive ruxolitinib phosphate PO BID on days 1-21 and paclitaxel and carboplatin as in arm I. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Within 6 weeks after completion of cycle 3, patients undergo TRS.

ARM II (CYCLES 4-6): Within 4 weeks of surgery (or within 6 weeks of completion of cycle 3 in patients who do not undergo TRS), patients receive ruxolitinib phosphate PO BID on days 1-21 and paclitaxel and carboplatin as in arm I. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients in phase I are followed up until resolution of adverse events, and patients in phase II are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinically and radiographically suspected and previously untreated International Federation of Gynecologic and Obstetrics (FIGO) stage III or IV epithelial ovarian, primary peritoneal or fallopian tube cancer, high grade, for whom the plan of management will include neoadjuvant chemotherapy (NACT) with interval tumor reductive surgery (TRS) who have undergone biopsies for histologic confirmation
* Institutional confirmation of Mullerian epithelial adenocarcinoma on core biopsy (not cytology or fine needle aspiration) or laparoscopic biopsy; (for phase II of the study formalin-fixed paraffin-embedded [FFPE] tissue should be available for laboratory analysis); patients with the following histologic epithelial cell types are eligible: high grade serous carcinoma, high grade endometrioid carcinoma, clear cell carcinoma, or a combination of these
* All patients must have measurable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination within 28 days prior to registration
  * Radiographic imaging of the chest, abdomen and pelvis within 28 days prior to registration documenting disease consistent with FIGO stage III or IV disease
  * Further protocol-specific assessments
* Eastern Cooperative Oncology Group (ECOG)/Karnofsky performance status of 0, 1, or 2 within 28 days prior to registration
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl; this ANC cannot have been induced by granulocyte colony stimulating factors (within 14 days prior to registration)
* Platelets greater than or equal to 100,000/mcl (within 14 days prior to registration)
* Hemoglobin greater than 9.0 mg/dl (transfusions are permitted to achieve baseline hemoglobin level) (within 14 days prior to registration)
* Estimated creatinine clearance (CrCl) >= 50 mL/min according to the Cockcroft-Gault formula (within 14 days prior to registration)
* Bilirubin =< 1.5 x upper limit of normal (ULN) (within 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (within 14 days prior to registration)
* Alkaline phosphatase =< 2.5 x ULN (within 14 days prior to registration)
* Neurologic function: neuropathy (sensory and motor) less than or equal to Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Ability to swallow and retain oral medication
* The patient must provide study-specific informed consent prior to study entry
* BRCA testing results (i.e., comprehensive BRCA1 and BRCA2 sequencing, including assessment of gene rearrangements) must be submitted for all patients enrolled to Amendment 7 and subsequent amendments; BRCA testing results are optional for all patients enrolled prior to Amendment 7; due to the long acceptance of germline BRCA testing through Myriad, Myriad testing reports will be accepted without additional documentation; if testing for germline BRCA is done by other organizations, in addition to the testing report, documentation from a qualified medical professional (e.g., ovarian cancer specialty physician involved in the field, high risk genetics physician, genetics counselor) detailing the laboratory results is required; please retain a copy of all reports (positive, variants of unknown significance [VUS], or negative)

Exclusion Criteria:

* Patients with suspected non-gynecologic malignancy, such as gastrointestinal
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies are excluded if there is any evidence of other malignancy being present within the last three years (2 years for breast cancer); patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor within the last three years are excluded; patients may have received prior adjuvant chemotherapy and radiotherapy for localized breast cancer, provided that it was completed more than 2 years prior to registration, the patient remains free of recurrent or metastatic disease and hormonal therapy has been discontinued
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis or thoracic cavity within the last three years are excluded; prior radiation for localized cancer of the head and neck or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received any targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management of their epithelial ovarian, fallopian tube or peritoneal primary cancer
* Patients with mucinous carcinoma, low grade endometrioid carcinoma, low grade serous carcinoma or carcinosarcoma
* Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, unless all of the following conditions are met: stage not greater than I-A, grade 1 or 2, no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including serous, clear cell or other FIGO grade 3 lesions
* Severe, active co-morbidity defined as follows:

  * Chronic or current active infectious disease requiring systemic antibiotics, antifungal or antiviral treatment
  * Known brain or central nervous system metastases or history of uncontrolled seizures
  * Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months from enrollment, New York Heart Association class III or IV congestive heart failure, and serious arrhythmia requiring medication (this does not include asymptomatic atrial fibrillation with controlled ventricular rate)
  * Partial or complete gastrointestinal obstruction
* Patients who are not candidates for major abdominal surgery due to known medical comorbidities
* Patients with any condition that in the judgment of the investigator would jeopardize safety or patient compliance with the protocol
* Patients who are unwilling to be transfused with blood components
* Concurrent anticancer therapy (e.g. chemotherapy, radiation therapy, biologic therapy, immunotherapy, hormonal therapy, investigational therapy)
* Receipt of an investigational study drug for any indication within 30 days or 5 half-lives (whichever is longer) prior to day 1 of protocol therapy
* Patients who, in the opinion of the investigator, are unable or unlikely to comply with the dosing schedule and study evaluations
* Patients who are pregnant or nursing; the effects of ruxolitinib on the developing human fetus are unknown; for this reason, women of child-bearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; WOCBP must have a screening negative serum or urine pregnancy test within 14 days of registration; a second pregnancy test must be done within 24 hours prior to the start of the first cycle of study treatment; women must not be breastfeeding

  * Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) do not require contraception
  * Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy and/or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 month amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level greater than 40mIU/mL
* Known history of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection or known history of tuberculosis; (This exclusion criterion is necessary because the treatments involved in this protocol may be immunosuppressive)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles N Landen, Principal Investigator — NRG Oncology
Locations (110):
- United States (110):
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Sutter Auburn Faith Hospital, Auburn, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Danbury Hospital, Danbury, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Women's Cancer Care-Covington, Covington, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

REFERENCES:
- [Derived] Landen CN, Buckanovich RJ, Sill MW, Mannel RS, Walker JL, DiSilvestro PA, Mathews CA, Mutch DG, Hernandez ML, Martin LP, Bishop E, Gill SE, Gordinier ME, Burger RA, Aghajanian C, Liu JF, Moore KN, Bookman MA. Phase I and Randomized Phase II Study of Ruxolitinib With Frontline Neoadjuvant Therapy in Advanced Ovarian Cancer: An NRG Oncology Group Study. J Clin Oncol. 2024 Jul 20;42(21):2537-2545. doi: 10.1200/JCO.23.02076. Epub 2024 May 22. PMID 38776484

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2 - Arm I (Paclitaxel and Carboplatin): See Detailed Description.
  Carboplatin: Given IV
  Paclitaxel: Given IV
  Therapeutic Conventional Surgery: Undergo TRS
- Phase 2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin): See Detailed Description.
  Carboplatin: Given IV
  Paclitaxel: Given IV
  Ruxolitinib Phosphate: Given PO
  Therapeutic Conventional Surgery: Undergo TRS
- Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin): See Detailed Description.
  Carboplatin: Given IV (AUC 5)
  Paclitaxel: Given IV (70 mg/m2/week)
  Ruxolitinib Phosphate: Given PO (15 mg bid)
- Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin): See Detailed Description.
  Carboplatin: Given IV (AUC 6)
  Paclitaxel: Given IV (70 mg/m2/week)
  Ruxolitinib Phosphate: Given PO (10 mg bid)
Period: Phase 1 - Dose Level 1
Arm/Group | Phase 2 - Arm I (Paclitaxel and Carboplatin) | Phase 2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Started | 0 | 0 | 7 | 0
Completed | 0 | 0 | 7 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase 1 - Dose Level 2
Arm/Group | Phase 2 - Arm I (Paclitaxel and Carboplatin) | Phase 2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Started | 0 | 0 | 0 | 10
Completed | 0 | 0 | 0 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 2 - Arm I (Paclitaxel and Carboplatin) | Phase 2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Started | 42 | 88 | 0 | 0
Completed | 42 | 88 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable
Groups:
- Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin); Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin): See Detailed Description.
  Carboplatin: Given IV
  Paclitaxel: Given IV
  Ruxolitinib Phosphate: Given PO
  Therapeutic Conventional Surgery: Undergo TRS
- Total: Total of all reporting groups
Arm/Group | Phase 2 - Arm I (Paclitaxel and Carboplatin) | Phase 2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Total
Number analyzed (Participants) | 42 | 88 | 7 | 10 | 147
Age, Customized [Count of Participants; unit: Participants]
  20 - 29 years | 0 | 0 | 0 | 0 | 0
  30 - 39 years | 2 | 2 | 1 | 1 | 6
  40 - 49 years | 1 | 6 | 0 | 1 | 8
  50 - 59 years | 6 | 19 | 1 | 2 | 28
  60 - 69 years | 11 | 30 | 3 | 3 | 47
  70 - 79 years | 22 | 27 | 2 | 3 | 54
  >= 80 years | 0 | 4 | 0 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 88 | 7 | 10 | 147
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 0 | 1 | 12
  Not Hispanic or Latino | 34 | 79 | 7 | 9 | 129
  Unknown or Not Reported | 2 | 4 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 0 | 0 | 7
  White | 38 | 80 | 6 | 9 | 133
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities (Phase I)
Description: Will be assessed according to Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 (CTCAE version 5.0 will be used starting 04/01/2018), or delays in treatment caused by toxicities. A DLT is defined as either hematologic or non-hematologic toxicity (assessed in accordance with the CTEP CTCAE Version 4.0), which cause any of the following (any toxicity): a dose delay > 7 days related to any toxicity, an omission of day 8 or day 15 paclitaxel, any treatment related death. For hematologic toxicity: study treatment-related febrile neutropenia, grade 4 neutropenia lasting > 7 days, study treatment-related grade 4 thrombocytopenia or bleeding associated with grade 3 thrombocytopenia. For non-hematologic toxicity: study treatment related grade 3 or grade 4 non-hematologic toxicity.
Time Frame: 42 days (2 cycles)
Population: Eligible
Measure: Number; unit: participants
Arm/Group | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Number analyzed (Participants) | 7 | 7
participants | 2 | 3

2. Primary Outcome: Progression-free Survival (PFS) (Phase II)
Description: Will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. A log-rank test utilizing the categorized values of the exploratory laboratory parameters or a Cox proportional hazards (PH) model to estimate of the hazard ratio for progression or death in PFS. If feasible, the PH model will examine the effect of continuous measures.
  All patients must have measurable disease, and at least one "target lesion" to be used to assess response as defined by RECIST 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray. Lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
Time Frame: The maximum follow-up time for PFS is 57 months.
Population: Eligible for PFS analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 - Arm I (Paclitaxel and Carboplatin) | Phase 2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Number analyzed (Participants) | 42 | 88
months | 11.63 [10.32 to 14.39] | 14.55 [11.89 to 16.92]

3. Secondary Outcome: Number of Participants With Grade 3 or Higher AE (Phase I and II)
Description: Will be assessed according to CTEP CTCAE version 4.03 (CTCAE version 5.0 will be used starting 04/01/2018). Count of Participants with grade 3 or higher AE. The participants included are the patients in Arm I and the patients in Arm II (DL1 and phase 2). The patients in phase 1 DL2 are not included because they are at a different dose level.
  The first 17 patients were entered between 11/14/2016 and 10/19/2017. These are the phase 1 patients. Group in DL1 entered 7 patients between 11/14/2016 - 2/17/2017. The DL2 patients were entered between 4/21/2017 and 10/19/2017. There were 10 entered in DL2 because we had a few (3 patients) who were not evaluable and needed to be replaced. From 6/28/2018 to 2/3/2020, we entered the phase 2 patients (42 vs. 88). The first 7 patients were combined with the active therapy on phase 2, for the toxicity comparison (42 vs. 88+7=95 patients).
Time Frame: Serious and other adverse events were collected from baseline until 30 days after last treatment, an average of 10 months.
Population: Eligible
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 - Arm I (Paclitaxel and Carboplatin) | Phase 2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Number analyzed (Participants) | 42 | 88 | 7 | 10
Participants | 32 | 81 | 1 | 3

4. Secondary Outcome: Frequency of Patients Who Could Not Receive Surgery Within the Defined Timeframe for Reasons Other Than Non-response, Disease Progression, or Medical Contraindications (Phase I)
Description: Frequencies will be given by the dose-level administered.
Time Frame: Up to 6 weeks
Population: Eligible
Measure: Number; unit: participants
Arm/Group | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Number analyzed (Participants) | 7 | 10
participants | 0 | 3

5. Secondary Outcome: Number of Patients Who Discontinue Ruxolitinib in the First 3 Months of Maintenance Therapy Due to Toxicity (Phase I)
Description: Number of patients who discontinue ruxolitinib in the first 3 months of maintenance therapy due to toxicity (Phase I)
Time Frame: Up to 3 months in the maintenance phase
Population: Eligible
Measure: Number; unit: participants
Groups:
- Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel and Carboplatin); Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin): See Detailed Description.
  Carboplatin: Given IV
  Paclitaxel: Given IV
  Ruxolitinib Phosphate: Given PO
  Therapeutic Conventional Surgery: Undergo TRS
Arm/Group | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel and Carboplatin) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

6. Secondary Outcome: Progression-free Survival (PFS) (Phase II) (Subset Analysis)
Description: Will be assessed according to RECIST 1.1. Subset analyses within categorized, important exploratory laboratory parameters will examine the treatment effect on PFS. The effect of treatment on PFS will be examined within each of these subsets using a log-rank test or a Cox PH model. Interest will center on whether the hazard of PFS changes from one group to another. The impact of the biomarkers on PFS will be assessed using log-rank tests or Cox PH models.
Time Frame: From study entry to time of progression or death, whichever occurs first, assessed up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-03

7. Secondary Outcome: Number of Patients Who Have Total Gross Resection (Phase II)
Description: The outcome is whether there is a total gross resection rate at time of interval cytoreductive surgery among those who had surgery.
Time Frame: At the time of surgery (surgery occurred within 6 weeks after completion of cycle 3, as soon as nadir counts permit and surgery deemed safe by investigator)
Population: Eligible
Measure: Number; unit: participants
Arm/Group | Arm I (Paclitaxel and Carboplatin) | Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Number analyzed (Participants) | 35 | 77
participants | 20 | 49

8. Secondary Outcome: Number of Participants With Complete Pathological Response (Phase II)
Description: At the time of TRS, complete pathologic response is defined as no evidence of disease on radiographic imaging at the time of radiographic tumor measurement just prior to TRS, no visible or palpable tumor at the time of surgical exploration, and no pathologic evidence of disease in tissue specimens obtained from TRS.
Time Frame: At the time of tumor reductive surgery or biopsy after 3 cycles (i.e. after 63 days).
Population: Eligible
Measure: Number; unit: participants
Arm/Group | Arm I (Paclitaxel and Carboplatin) | Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Number analyzed (Participants) | 35 | 77
participants | 0 | 1

9. Secondary Outcome: Overall Survival (OS) (Phase II)
Description: The effect of treatment on OS will be conducted with a Kaplan-Meier analysis and reported as median survival times.
Time Frame: The average (median) OS follow-up time is 38 months.
Population: Eligible
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel and Carboplatin) | Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
Number analyzed (Participants) | 42 | 88
months | 30.8 [24.6 to NA] — Due to insufficient sample size, lack of follow-up time or a lack of a sufficient probability of death, the upper limit of the 95% CI for Arm I is not able to be estimated (NA). | NA [30.9 to NA] — Due to insufficient sample size, lack of follow-up time or a lack of a sufficient probability of death, the median and upper limit of the 95% CI for Arm II is not able to be estimated (NA).

10. Other Pre Specified Outcome: Change in Cancer Stem Cells (CSC) Observed in Tissue
Description: Landmark analyses will be conducted to see if changes in CSC are associated with PFS. The predictive value of CSC will be formally examined with a Cox model using an interaction term with treatment. Subset analyses will be conducted as well in the event that a formal analysis fails to reject the null hypothesis.
Time Frame: Baseline up to 63 days (3 cycles)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Serum C-reactive Protein (CRP)
Description: The impact of baseline values on PFS and OS can be assessed for prognostic and predictive significance with log-rank statistics and Cox models. The impact of changes in CRP values on PFS and OS can be examined with landmark analyses or as time dependent covariates.
Time Frame: Baseline up to 63 days (3 cycles)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were collected from baseline until 30 days after the last treatment, an average of 10 months. All-Cause Mortality was collected from baseline until end of follow-up, an average of 38 months.
Description: Will be assessed according to CTEP CTCAE version 4.03 (CTCAE version 5.0 will be used starting 04/01/2018).
Arm/Group | Phase 2 - Arm I (Paclitaxel and Carboplatin) | Phase 2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin)
All-Cause Mortality (participants affected / at risk) | 14/42 | 25/88 | 4/7 | 10/10
Serious Adverse Events (participants affected / at risk) | 9/42 | 42/88 | 1/7 | 3/10
Other Adverse Events (participants affected / at risk) | 41/42 | 88/88 | 1/7 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2 - Arm I (Paclitaxel and Carboplatin) (N=42) | Phase 2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) (N=88) | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) (N=7) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) (N=10)
Anemia (Blood and lymphatic system disorders) | 2 | 15 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 6 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 8 | 0 | 1
Death NOS (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 3 | 0 | 0
Sepsis (Infections and infestations) | 0 | 4 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 0
Wound infection (Infections and infestations) | 0 | 3 | 0 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cardiac troponin I increased (Investigations) | 1 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 10 | 0 | 0
Platelet count decreased (Investigations) | 2 | 3 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 4 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucinations (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 8 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2 - Arm I (Paclitaxel and Carboplatin) (N=42) | Phase 2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) (N=88) | Phase 1 - DL1 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) (N=7) | Phase 1 - DL2 - Arm II (Ruxolitinib, Paclitaxel, and Carboplatin) (N=10)
Anemia (Blood and lymphatic system disorders) | 28 | 70 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 6 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 7 | 7 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 3 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Blurred vision (Eye disorders) | 1 | 4 | 0 | 0
Dry eye (Eye disorders) | 0 | 2 | 0 | 0
Eyelid function disorder (Eye disorders) | 0 | 1 | 0 | 0
Flashing lights (Eye disorders) | 0 | 1 | 0 | 0
Periorbital edema (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 9 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 16 | 44 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 5 | 0 | 0
Bloating (Gastrointestinal disorders) | 8 | 7 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 17 | 41 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 20 | 40 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 4 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 6 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 5 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 7 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 5 | 22 | 0 | 0
Nausea (Gastrointestinal disorders) | 24 | 51 | 0 | 1
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatic fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 11 | 30 | 0 | 1
Chills (General disorders) | 1 | 3 | 0 | 0
Death NOS (General disorders) | 1 | 0 | 0 | 0
Edema face (General disorders) | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 10 | 18 | 0 | 0
Fatigue (General disorders) | 30 | 63 | 0 | 1
Fever (General disorders) | 1 | 9 | 0 | 0
Flu like symptoms (General disorders) | 0 | 3 | 0 | 0
Localized edema (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 3 | 0 | 0
Neck edema (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 7 | 0 | 0
Pain (General disorders) | 6 | 7 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 1 | 0 | 0
Bladder infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 2 | 0 | 0
Eye infection (Infections and infestations) | 1 | 2 | 0 | 0
Lung infection (Infections and infestations) | 2 | 6 | 0 | 0
Otitis media (Infections and infestations) | 0 | 2 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 4 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 3 | 3 | 0 | 0
Upper respiratory infection (Infections and infestations) | 2 | 7 | 0 | 0
Urinary tract infection (Infections and infestations) | 6 | 12 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 2 | 0 | 0
Wound infection (Infections and infestations) | 3 | 4 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 3 | 12 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 7 | 0 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 7 | 16 | 0 | 0
Alkaline phosphatase increased (Investigations) | 7 | 12 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 7 | 12 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0
Cardiac troponin I increased (Investigations) | 1 | 0 | 0 | 0
Creatinine increased (Investigations) | 3 | 10 | 0 | 0
INR increased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 9 | 16 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 22 | 63 | 0 | 0
Platelet count decreased (Investigations) | 16 | 40 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0
Weight gain (Investigations) | 2 | 2 | 0 | 0
Weight loss (Investigations) | 10 | 16 | 0 | 0
White blood cell decreased (Investigations) | 19 | 36 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 8 | 17 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 10 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 14 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 | 19 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 15 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 17 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 26 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 9 | 15 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 10 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 | 6 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 7 | 0 | 0
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 14 | 22 | 1 | 0
Dysgeusia (Nervous system disorders) | 8 | 18 | 0 | 0
Headache (Nervous system disorders) | 6 | 19 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 2 | 0 | 0
Paresthesia (Nervous system disorders) | 2 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 20 | 40 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 7 | 10 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 7 | 0 | 0
Hallucinations (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 8 | 13 | 0 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 2 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 5 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 3 | 5 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 5 | 6 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 2 | 0 | 0 | 0
Genital edema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 4 | 0 | 0
Vaginal fistula (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 3 | 7 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 18 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 | 29 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 23 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 48 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 6 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 8 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 3 | 0 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hot flashes (Vascular disorders) | 2 | 9 | 0 | 0
Hypertension (Vascular disorders) | 9 | 19 | 0 | 0
Hypotension (Vascular disorders) | 5 | 11 | 1 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischemia (Vascular disorders) | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 15 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT02713386/Prot_SAP_000.pdf